CLINICAL TRIAL: NCT03896841
Title: Ocular Surface Disease Test Results, Corneal Biomechanical Properties, and Structural Parameters in Patients With Polycystic Ovary Syndrome
Brief Title: Ocular Findings of Polycystic Ovary Syndrome
Status: Completed | Type: Observational
Sponsor: Istanbul Medeniyet University (Other)
Responsible Party: Principal Investigator, Mustafa Hepokur, Medical Doctor, Clinical Investigator, Istanbul Medeniyet University
Other Study IDs: 25801608
Record Dates: First submitted 2019-01-13; First posted 2019-04-01 (Actual); Last update posted 2019-04-01 (Actual); Status verified 2019-01

CONDITIONS: Polycystic Ovary Syndrome
MeSH Terms: conditions — Polycystic Ovary Syndrome | interventions — Observation

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- PCOS: premenopausal patients with PCOS
  Interventions: Other: Observation
- control subjects: non-pregnant healthy control subjects
  Interventions: Other: Observation

INTERVENTIONS:
Other: Observation — Ocular Findings Observations

SUMMARY:
Purpose: This study aimed to compare the ocular surface disease test results, anterior segment parameters, and ocular response analyzer (ORA) findings of polycystic ovary syndrome (PCOS) patients with those of healthy reproductive age female controls.

ELIGIBILITY:
Inclusion Criteria:

* premenopausal with PCOS

Exclusion Criteria:

* patients with external ocular disease other than dry eye complaints,
* use of topical drops that can affect the tear film layer,
* contact lens use histories,
* those who received hormone therapy for 6 months,
* those who have systemic medication or systemic disease that may affect the tear film layer and reproductive physiology,
* previous eye surgeries,
* smokers and alcohol users,
* those having diseases (Cushing's syndrome or androgen-secreting tumors) causing similar clinical findings.

Ages: 19 Years to 43 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: This was a prospective, case-control study in which 23 premenopausal patients with PCOS diagnoses and 15 non-pregnant healthy control subjects were included.
Sampling Method: Probability Sample
Enrollment: 38 (Actual)
Dates: Start 2013-03-17 (Actual); Primary Completion 2014-03-20 (Actual); Study Completion 2018-03-30 (Actual)

PRIMARY OUTCOMES:
Comparison of the anterior segment parameter results (Pentacam). | 1 year
  measurement of the central corneal thickness.
Comparison of the corneal biomechanical parameter results (ocular response analyzer). | 1 year
  measurement of the corneal hysteresis (CH).

IPD SHARING:
Plan to Share IPD: No